CLINICAL TRIAL: NCT02546440
Title: Phase IIA Study on Therapy With the NF-κB Inhibiting and Apoptosis Inducing Drug Dimethylfumarate (DMF) in Patients With Cutaneous T Cell Lymphoma (CTCL)
Brief Title: Study on Therapy With Dimethylfumarate (DMF) in Patients With Cutaneous T Cell Lymphoma (CTCL)
Acronym: DMF-CTCL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitätsmedizin Mannheim (Other)
Collaborators: Klinikum Minden (Unknown); Klinikum Krefeld (Unknown); Wuerzburg University Hospital (Other); KKS Netzwerk (Network); Klinikum Ludwigshafen (Other); Universitätsklinikum Kiel (Unknown)
Responsible Party: Principal Investigator, Jan Nicolay, MD MSc, Universitätsmedizin Mannheim
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT-Number: 2014-000924-11
Record Dates: First submitted 2015-09-06; First posted 2015-09-10 (Estimated); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Cutaneous T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous | interventions — Dimethyl Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- treatment arm (Experimental): patients are treated with dimethylfumarate over 24 weeks. Dosage will be escalated weekly from 30 mg/d to 720 mg/d over 9 weeks. The dose escalation scheme is the same as approved for psoriasis treatment in Germany
  Interventions: Drug: Dimethyl fumarate

INTERVENTIONS:
Drug: Dimethyl fumarate — dose escalation from 30 mg/d to maximally 720 mg/d over 9 weeks, then continuing with the highest tolerated dose following a preset design in psoriasis treatment in Germany, oral medication in tablet form. Treatment will last 24 weeks or until either progression or unacceptable side effects occur

SUMMARY:
The main objective of the trial is to investigate whether oral treatment of patients suffering from cutaneous T cell lymphoma with dimethylfumarate is leading to a significant improvement of modified severity assessment tool (mSWAT) values in the skin after 24 weeks of treatment (primary endpoint). Secondary endpoints are dermatologic life quality index, itching and pain measured by a NRS and the blood involvement if applicable.

Primary: safety and efficacy of DMF treatment in CTCL Secondary: Dermatologic Life Quality index, NRS for itching and pain, blood involvement if appl.

ELIGIBILITY:
Inclusion criteria:

* Histopathologically confirmed Mycosis fungoides or Sézary syndrome (CTCL stage ≥ Ib according to EORTC-ISCL consensus classification) at study entry with progressive, persistant or recurrent disease
* Pretreatment with at least one topical or systemic CTCL therapy or UV therapy, if the prior therapy is not possible anymore or if there is new contraindication or unsatisfactory response
* Karnofsky index ≥70 % (according to Karnofsky DA, Burchenal JH. (1949). "The Clinical Evaluation of Chemotherapeutic Agents in Cancer." In: MacLeod CM (Ed), Evaluation of Chemotherapeutic Agents. Columbia Univ Press. Page 196)
* Life expectancy > 3 months
* Age ≥ 18 years
* Adequate organ function:
* differential blood count: hemoglobin ≥ 10 g/dl without transfusions, leukocyte count > 3000/µl, lymphocyte count > 700/µl
* liver enzymes ≤ 2 x upper limit of normal (ULN)
* serum creatinine ≤ 1.5 mg/dl or calculate creatinine clearance ≥ 50 ml/min,
* Negative Pregnancy test from blood, agreement for efficient contraception in male and female patients unless infertility is documented (DMF is not approved during pregnancy)
* Ability to understand character and individual consequences of the clinical trial and to provide written informed consent to participate in the study
* written informed consent must be given according to ICH/GCP, and national/local regulations, before patient registration and prior to any study specific procedures.

Exclusion criteria:

* Another active malignant disease with the following exceptions:
* Basal or squamous cell carcinoma of the skin
* In situ carcinoma of the cervix or the skin
* Topical chemotherapy, superficial radiotherapy, photopheresis or systemic CTCL treatment within 28 days before study therapy initiation
* Severe systemic disease or infection at study therapy initiation
* Prior treatment with DMF or simultaneous topical DMF treatment
* Contraindications for treatment with DMF (known hypersensibility to the drug, severe gastrointestinal disease (like ulcerations), Alcohol abuse, other obligately liver- or nephrotoxic medication, known clinically apparent renal or hepatic insufficiency)
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
* Participation in other clinical studies within 14 days before study therapy initiation
* Pregnant or lactating patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2021-09 (Actual); Study Completion 2022-09 (Actual)

PRIMARY OUTCOMES:
safety (via occurrence of AE/SAE) of DMF treatment in CTCL | every 2 weeks until 24 weeks of treatment are finished
  Number of patients with Treatment-related Adverse Events as assessed by CTCAE v4.0
efficacy (via improvement of Skin involvement measured by the standardized modified severity weighted assessment tool (mSWAT))of DMF treatment in CTCL | every 2 weeks until 24 weeks of treatment are finished
  Changes in the mSWAT scores range from 0 [no patches, Plaques or tumors on the Skin ] to 400 [complete Body covered by Tumors]

SECONDARY OUTCOMES:
changes in dermatologic life quality index | every 2 weeks until 24 weeks of treatment are finished
  Scores range from 0 [no restriction of life Quality] to 30 [maximal restriction of life Quality]
changes in pruritus intensity measured by a visual analog scale | every 2 weeks until 24 weeks of treatment are finished
  Scores range from 0 [no Pruritus] to 10 [worst possible Pruritus]
changes in blood involvement measured by Sezary cell count (if applicable, only in stage IV patients) | every 2 weeks until 24 weeks of treatment are finished

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center, Mannheim, Germany

REFERENCES:
- [Derived] Nicolay JP, Melchers S, Albrecht JD, Assaf C, Dippel E, Stadler R, Wehkamp U, Wobser M, Zhao J, Burghaus I, Schneider S, Gulow K, Goerdt S, Schurch CM, Utikal JS, Krammer PH. Dimethyl fumarate treatment in relapsed and refractory cutaneous T-cell lymphoma: a multicenter phase 2 study. Blood. 2023 Aug 31;142(9):794-805. doi: 10.1182/blood.2022018669. PMID 37217183